**abbyie** AGN-242428 and AGN-231868 2012-201-005 – Statistical Analysis Plan (Stage 2) Version 1.0 - 07 December 2021

## Statistical Analysis Plan for Study 2012-201-005 Stage 2

A Multicenter, Vehicle-controlled, Randomized Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of AGN-242428 and **AGN-231868** in Participants with Dry Eye Disease

Date: 07 December 2021

Version 1.0

## **Table of Contents**

| 1.0 | Introduction | 5 |
|---|---|---|
| 2.0 | Study Design and Objectives | |
| 2.1 | Objectives and Hypothesis | 5 |
| 2.2 | Study Design Overview | 6 |
| 2.3 | Treatment Assignment and Masking | 8 |
| 2.4 | Sample Size Determination | 9 |
| 3.0 | Endpoints | 9 |
| 3.1 | Safety Endpoints | 9 |
| 3.2 | Secondary endpoints | 10 |
| 3.3 | | 10 |
| 4.0 | Analysis Populations | |
| 5.0 | Subject Disposition | 12 |
| 6.0 | Study Drug Duration and Compliance | 13 |
| 7.0 | Demographics, Baseline Characteristics, Medical History, and Prior/Concomitant Medications | 13 |
| 7.1 | Demographics and Baseline Characteristics | 13 |
| 7.2 | Medical History | 13 |
| 7.3 | Prior and Concomitant Medications | 14 |
| 8.0 | Efficacy Analyses | 14 |
| 8.1 | General Considerations | 14 |
| 8.2 | Handling of Missing Data | 15 |
| 8.3 | | |
| 8.3.1 | | |
| 8.3.2 | | |
| 8.3.3 | | |
| 8.3.4 | | |
| 8.4 | | |
| 9.0 | Safety Analyses | 17 |
| 9.1 | General Considerations | 17 |
| 9.2 | Adverse Events | 18 |
| 9.2.1 | Treatment-Emergent Adverse Events | 18 |

# AGN-242428 and AGN-231868 2012-201-005 – Statistical Analysis Plan (Stage 2) Version 1.0 – 07 December 2021

| 9.2.2 | Adverse Event Overview | 19 |
|---|---|---|
| 9.2.3 | Treatment-Emergent Adverse Events by SOC and/or PT | |
| 9.2.4 | SAEs (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation | |
| 9.2.5 | Adverse Events of Special Interest | |
| 9.3 | Analysis of Laboratory Data | |
| 9.4 | Analysis of Vital Signs | 21 |
| 9.5 | Analysis of Electrocardiograms | 22 |
| 9.6 | Analysis of Best-corrected Visual Acuity | 22 |
| 9.7 | Intraocular Pressure | 22 |
| 9.8 | Biomicroscopy and Ophthalmoscopy | 22 |
| 9.9 | Safety Subgroup Analyses (if applicable) | 23 |
| 10.0 | Interim Analyses | 24 |
| 11.0 | Version History | 24 |
| 12.0 | Appendices | 24 |
| List of Table 1. | Stage 2 - Study Objectives and Assessments/Endpoints | 6 |
| Table 2. | | |
| Table 3. | Analysis Populations | |
| Table 4. | SAP Version History Summary | 24 |
| Table 5. | List of Preferred Terms for Adverse Events of Special Interest | 26 |
| Table 6. | Potentially Clinically Significant Criteria for Clinical Laboratory Parameters | 27 |
| Table 7. | Potentially Clinically Significant Criteria for Vital Signs Parameters | 28 |
| Table 8. | Potentially Clinically Significant Criteria for ECG Parameters | 29 |
| List of Fi | gures | |
| Figure 1. | | |



## **List of Appendices**

| Appendix A. | Protocol Deviations | 25 |
|---|---|---|
| Appendix B. | Definition of Adverse Events of Special Interest | 26 |
| Appendix C. | Potentially Clinically Significant Criteria for Safety Endpoints | 27 |
| Appendix D. | List of Abbreviations | 30 |
| Appendix E. | Changes to Protocol-planned Analyses | 31 |



#### 1.0 Introduction

This Statistical Analysis Plan (SAP) provides a technical and detailed elaboration of the statistical analyses of the efficacy and safety data for Stage 2 of this study as outlined and specified in the 2012-201-005 protocol amendment 3 (approved version dated 19 July 2021). Specifications of tables, figures and data listings are contained in a separate document. Details of the analyses of pharmacokinetic data will be documented separately before final database lock.

The SAP will not be updated in case of administrative changes or amendments to the protocol unless the changes impact the analysis.

Unless noted otherwise, all analyses will be performed using SAS Version 9.4 (SAS Institute Inc., Cary, NC 27513) or later under the Linux operating system.

#### 2.0 Study Design and Objectives

#### 2.1 Objectives and Hypothesis

This is the first-in-human study to evaluate the safety, tolerability, PK, and efficacy of AGN-242428 and AGN-231868 administered through topical ocular instillation. Data collected from animal studies suggest that both interventions have a good safety profile and the potential to reduce the signs and symptoms of dry eye disease (DED). Data from this study will guide future development of either or both compounds for the treatment of DED.



Table 1. Stage 2 - Study Objectives and Assessments/Endpoints

| Objectives | Assessments/Endpoints |
|---|---|
| Primary | |
| <ul> <li>To evaluate the safety and tolerability of<br/>AGN-242428 and AGN-231868 and their<br/>respective vehicles in participants with<br/>DED</li> </ul> | <ul> <li>AEs, clinical laboratory values, vital signs,<br/>ECG findings, IOP, BCVA, slit lamp<br/>biomicroscopy, dilated fundus examination,<br/>Drop Tolerability Questionnaire score</li> </ul> |
| Secondary | |
| <ul> <li>To assess the plasma exposure of<br/>AGN-242428 and AGN-231868; and tear<br/>exposure of AGN-242428, AGN-231868,<br/>and lifitegrast in participants with DED<br/>following twice daily dosing for up to<br/>6 weeks</li> </ul> | • Trough plasma or tear concentration ( $C_{trough}$ ) and plasma or tear concentration at 0.5 hours post-dose ( $C_{0.5h}$ ) |
| Tertiary/Exploratory | |

## 2.2 Study Design Overview

This is a Phase 1/2a, multicenter, vehicle-controlled, double-masked, randomized study conducted in 2 consecutive stages in participants with DED. Stage 1 was conducted at 2 sites in the United States and Stage 2 will be conducted at up to approximately 8 sites in the United States.



The Stage 2 schematic for the study is shown in Figure 1.

Figure 1. Study Schematic - Stage 2



## 2.3 Treatment Assignment and Masking

Participants will be randomized to one of the following study interventions in a 1:1:1:1:1 ratio:

- AGN-242428
- AGN-242428 vehicle
- AGN-231868

- AGN-231868 vehicle
- Xiidra



The AGN-242428, AGN-231868 and their vehicles will be provided in identical single-use vials. Xiidra will be supplied in single-use, commercially available vials that will have the original label overlaid with a new clinical label to prevent unmasking.

#### 2.4 Sample Size Determination

For Stages 1 and 2, the sample size is not based on statistical considerations and is determined empirically. Approximately 322 participants (72 in Stage 1 and 250 in Stage 2) will be enrolled in the study. No participant can be enrolled in more than 1 cohort and/or stage of the study.

## 3.0 Endpoints

## 3.1 Safety Endpoints

Safety endpoints are listed as the following:

AGN-242428 and AGN-231868 2012-201-005 – Statistical Analysis Plan (Stage 2) Version 1.0 – 07 December 2021

- adverse events (AEs),
- clinical laboratory values at the Exit/Early Termination visit,
- vital signs at each post-baseline visit,
- electrocardiogram (ECG) findings at the Exit/Early Termination visit,
- intraocular pressure (IOP) at each post-baseline visit,
- best-corrected visual acuity (BCVA) at each post-baseline visit,
- slit-lamp biomicroscopy findings at each post-baseline visit,
- dilated fundus (ophthalmoscopy) examination findings at the Exit/Early Termination visit.
- Drop Tolerability Questionnaire score at each post-baseline visit.

For eye-related endpoints, both eyes will be included in the analysis.

#### 3.2 Secondary endpoints

The secondary endpoints are trough plasma or tear concentration ( $C_{trough}$ ) and plasma or tear concentration at 0.5 hours post-dose ( $C_{0.5h}$ ). Details of endpoint and analysis will be included in a separate PK SAP.

#### 3.3 Tertiary/Exploratory Efficacy Endpoints



## 4.0 Analysis Populations

The analysis populations related to the statistical analysis detailed in this document will consist of participants as defined in Table 3. Additional analysis populations, such as PK population and biomarker population will be described separately in other analysis plans. There are a run-in period and a randomized study intervention period in Stage 2.

Table 3. Analysis Populations

| Population | Definition |
|---|---|
| Intent-to-Treat (ITT) | All participants who are randomized. Participants will be summarized according to the randomized study intervention. |
| Safety | All participants who receive $\geq 1$ administration of study intervention for Stage 2. |
| | <ul> <li>Safety population in randomized study intervention period includes<br/>all participants who receive ≥ 1 administration of randomized study<br/>intervention.</li> </ul> |
| | <ul> <li>The safety analysis will mainly be performed based on safety<br/>population in randomized study intervention period.</li> </ul> |
| | <ul> <li>Participants will be summarized according to the study drug that they<br/>actually received.</li> </ul> |
| | <ul> <li>Unless otherwise specified, study intervention and safety population<br/>will refer to the study intervention and safety population in<br/>randomized study intervention period in this SAP.</li> </ul> |

### 5.0 Subject Disposition

The number of participants who are screened and enter the run-in period for the study will be provided. The number of participants in the study populations (ITT population and Safety population) will be summarized by study intervention group.

The summary of study disposition post-randomization will be provided by study intervention group as randomized for the following:

- Number of participants randomized (this frequency count will be used as the denominator to calculate the percentages described below)
- Number and percentage of participants treated
- Number and percentage of participants completing the study
- Number and percentage of participants discontinued from the study
- Reasons for discontinuation from the study

In addition, a listing will be provided for participant disposition. A participant is counted as completing the study if he/she has completed all study visits including Day 42 (Exit)

Visit. Participants that exit the study prior to the Day 42 visit will be considered discontinued from the study.

#### 6.0 Study Drug Duration and Compliance

The exposure to study intervention, calculated as (last study intervention date - first study intervention date + 1), will be summarized using descriptive statistics by study intervention for the Safety population.

## 7.0 Demographics, Baseline Characteristics, Medical History, and Prior/Concomitant Medications

#### 7.1 Demographics and Baseline Characteristics

Demographic parameters (age [years]; sex; race; ethnicity) will be summarized descriptively by study intervention group for the ITT population.

Baseline characteristics including BCVA, IOP values and

weight, height, and body mass index will be summarized descriptively by study intervention group for the ITT population.

#### 7.2 Medical History

Medical history including prior procedures data will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 24.1 or higher. The actual version of the MedDRA coding dictionary will be noted in the statistical tables and clinical study report.

The number and percentage of participants in each medical history category (by MedDRA primary system organ class and preferred term) will be summarized. The system organ class (SOC) will be presented in alphabetical order, and the preferred terms will be presented in alphabetical order within each SOC. Participants reporting more than one condition/diagnosis will be counted only once in each row (SOC or preferred term).



An ophthalmic history will be determined as indicated on the Medical History form of eCRF (marked "OD," "OS," or "OU" to the question of "What was the location of the medical history condition/event?"). The ophthalmic medical history will be summarized in a similar way to medical history.

#### 7.3 Prior and Concomitant Medications

Medication terms will be coded using the World Health Organization (WHO) Drug Dictionary (Version WHODDMAR21B3G). The version of the dictionary will be noted in the statistical tables and clinical study report.

A prior medication is defined as any medication taken prior to the date of the first dose of study intervention. A concomitant medication is defined as any medication that starts prior to the date of the first dose of study intervention and continues to be taken after the first dose of study intervention or any medication that starts on or after the date of the first dose of study intervention.

The number and percentage of participants taking medications will be summarized by preferred drug name based on the World Health Organization (WHO) Drug Dictionary for both prior and concomitant medications, respectively.









## 8.4 Efficacy Subgroup Analyses

No subgroup analyses are planned.

## 9.0 Safety Analyses

#### 9.1 General Considerations

The below general considerations will be applied to safety analyses, unless specified otherwise.

• Safety analyses will be based on safety data using the safety population based on the actual treatment received.

- A participant's actual treatment will be determined by the first dose of study drug.
- In general, baseline is defined as the last non-missing scheduled assessment prior to the first administration of study intervention (non-missing assessment before Day 1 study intervention).
- The change from baseline values at a visit will be computed as the value for the post baseline visit minus the baseline value, unless otherwise indicated.
- Descriptive statistics for continuous variables include the sample size (n, mean, standard deviation, median, 1st and 3rd quartiles, minimum, and maximum).
- Summary statistics for categorical variables include the sample size (n), frequency count, and percentage.
- AEs and findings from biomicroscopy and ophthalmoscopy examinations will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 24.1 or higher, according to the version of the MedDRA coding dictionary used for the study at the time of database lock.

#### 9.2 Adverse Events

AEs will be summarized and presented using primary MedDRA SOCs and preferred terms (PTs). Specific adverse events will be counted once for each participant for calculating percentages, unless stated otherwise. In addition, if the same adverse event occurs multiple times for a participant, the highest severity and level of relationship to investigational product will be reported.

#### 9.2.1 Treatment-Emergent Adverse Events

An AE will be considered a treatment-emergent adverse event (TEAE) if the AE began or worsened (increased in severity or became serious) on or after the date of the first dose of study drug. Events where the onset date is the same as the study drug start date are assumed to be treatment emergent.

In general, the number and percentage of participants experiencing TEAEs will be summarized overall, as well as by primary MedDRA SOC and PT. The SOCs will be



presented in alphabetical order, and the PTs will be presented in decreasing frequency order on active study drug within each SOC. The number and percentage of participants experiencing TEAEs will also be summarized by PT for identifying common AEs. TEAEs by PT summaries will be presented in decreasing frequency order on active study drug.

#### 9.2.2 Adverse Event Overview

Adverse events will be classified into ocular AEs and non-ocular AEs. An ocular AE will be determined as indicated on the AE form of eCRF (marked "OD" or "OS" to the question of "what was the location of the adverse event?"), and thus are not limited to AEs with primary SOCs of eye disorders.

An overview of AEs will be presented consisting of the number and percentage of participants experiencing at least one event for each of the following AE categories:

- TEAEs
  - Ocular TEAEs
  - Non-ocular TEAEs
- TEAEs related to study drug
  - Ocular TEAEs related to study drug according to the investigator
  - Non-ocular TEAEs related to study drug according to the investigator
- Severe TEAEs
- Serious TEAEs
  - Ocular serious TEAEs
  - Non-ocular serious TEAEs
- TEAEs leading to withdrawal of study treatment
  - Ocular leading to withdrawal of study treatment
  - Non-ocular leading to withdrawal of study treatment
- TEAEs of special interest
- TEAEs leading to death

- All deaths
- COVID-19 infection.

#### 9.2.3 Treatment-Emergent Adverse Events by SOC and/or PT

Treatment-emergent adverse events will be summarized for each of the following AE categories:

- TEAEs by SOC and PT
  - Ocular TEAEs by SOC and PT
  - Non-ocular TEAEs by SOC and PT
- TEAEs by PT
- TEAEs related to study drug by SOC and PT
  - Ocular TEAEs related to study drug by SOC and PT
  - Non-ocular TEAEs related to study drug by SOC and PT
- TEAEs by SOC, PT, and maximum severity
  - Ocular TEAEs by SOC, PT, and maximum severity
  - Non-ocular TEAEs by SOC, PT, and maximum severity

Specific adverse events will be counted once for each participant for calculating percentages, unless stated otherwise.

If the same adverse event occurs multiple times for a participant, the highest severity and level of relationship to investigational product will be reported.

## 9.2.4 SAEs (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation

SAEs (including deaths) and AEs leading to study drug discontinuation will be summarized by SOC and PT and in listing format.



#### 9.2.5 Adverse Events of Special Interest

Summary table by PT will be provided for Adverse Events of Special Interest (AESI) as defined in Appendix B, which will also be provided in a listing.

#### 9.3 Analysis of Laboratory Data

Descriptive statistics for values and changes from the baseline in standard units at each assessment time point will be presented by study intervention group.

Clinical laboratory test values will be considered potentially clinically significant (PCS) if they meet either the lower-limit or upper-limit PCS criteria listed in Appendix C. The number and percentage of participants who have PCS post-baseline clinical laboratory values will be tabulated by study intervention for all scheduled postbaseline visit. The percentages will be calculated relative to the number of participants who have available non-PCS baseline values and at least 1 postbaseline assessment. The numerator will be the total number of participants with at least 1 PCS postbaseline value.

#### 9.4 Analysis of Vital Signs

Descriptive statistics for vital signs (systolic and diastolic blood pressure, pulse rate, weight, respiration rate, and temperature) and their changes from baseline at each assessment timepoint will be presented by study intervention group.

Selected vital signs will be considered potentially clinically significant (PCS) if they meet either the lower-limit or upper-limit PCS criteria listed in Appendix C. The number and percentage of participants who have PCS postbaseline vital sign values will be tabulated by study intervention for each postbaseline visit assessments. The percentages will be calculated relative to the number of participants who have available baseline values for those parameters with the change from baseline value criterion or non-PCS baseline values for those vital sign parameters without the change from baseline value criterion and at least 1 postbaseline assessment. The numerator will be the total number of participants with at least 1 PCS postbaseline value.

#### 9.5 Analysis of Electrocardiograms

Descriptive statistics for ECG parameters (heart rate, PR interval, QRS duration, QT interval, and QTc) at baseline, Exit visit (pre-CAE and post-CAE) or Early Termination visit, and changes from baseline at the Exit visit will be presented by study intervention group.

ECG values will be considered potentially clinically significant (PCS) if they meet either the lower-limit or upper-limit PCS criteria listed in Appendix C. The number and percentage of participants who have PCS postbaseline ECG values will be tabulated by study intervention for Exit visit (pre-CAE and post-CAE) and Early Termination visit assessments. The percentages will be calculated relative to the number of participants who have available non-PCS baseline values and at least 1 postbaseline assessment. The numerator will be the total number of participants with at least 1 PCS postbaseline value.

#### 9.6 Analysis of Best-corrected Visual Acuity

BCVA will be quantified using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity protocol. Descriptive statistics for BCVA and changes from baseline at each post-baseline visit will be presented by study intervention, and by study eye and nonstudy eye. Change from baseline will also be summarized by study intervention for each eye at each visit in a categorical tabulation as severe ( $\geq$  30 letters decrease from baseline), moderate ( $\geq$  15 and < 30 letters decrease from baseline) and no loss or mild (< 15 letters decrease from baseline).

#### 9.7 Intraocular Pressure

Descriptive statistics for IOP and changes from baseline at each post-baseline visit will be presented by study intervention for each eye.

#### 9.8 Biomicroscopy and Ophthalmoscopy

Biomicroscopy will be performed in each eye at each visit, by slit-lamp examination, without pupil dilation, including but not limited to lids/lashes, conjunctiva, cornea, and

anterior chamber. Observations for the examination will be graded on a 5-point scale (0=none, 0.5=trace, 1=mild, 2=moderate, 3=severe) except for a) the anterior chamber cells: 0=0 cells, +0.5=1-5 cells, +1=6-15 cells, +2=16-25 cells, +3=26-50 cells, and +4=> 50 cells; and b) flare: 0=none, +1=faint, +2=moderate, +3= marked and +4=intense).

will be summarized using descriptive statistics at all post-baseline visits and pre-/post-CAE when applicable. For Pre-CAE change from baseline, the Day 1 Pre-CAE value prior to the administration of the first administration of study intervention will be used as baseline. For Post-CAE change from baseline, the Day 1 Post-CAE value prior to the administration of the first administration of study intervention will be used as baseline.

The number of participants with biomicroscopy findings of ≥ 2-grade severity increase from baseline will be generated for MedDRA preferred terms recorded on the Ocular Biomicroscopic Exam eCRFs at each post-baseline visit by study intervention for each eye. For findings under other pathology which are not associated with a severity grade, a status change from absent to present will be treated as a 2-grade increase in the analysis. At least 2-grade increase in severity from baseline is defined as a change from no finding to 2 and above, from 0.5 to 2 and above, or from 1 to 3 and above from baseline at any of the follow-up visits. The number and percentage of participants with clinically significant biomicroscopy findings (at least 2-grade increase in severity from baseline) will be tabulated by finding category, and study intervention group.

The ophthalmoscopy findings will be summarized similarly.

## 9.9 Safety Subgroup Analyses (if applicable)

No safety subgroup analyses are planned.

## 10.0 Interim Analyses

An interim database lock occurred after completion of Stage 1, and the unmasking and data analyses were performed. This doesn't affect masking of Stage 2. At the end of study, the final database lock will occur.

## 11.0 Version History

Table 4.SAP Version History Summary

| Version | Date | Summary |
|---------|------------------|------------------|
| 1.0 | 07 December 2021 | Original version |

## 12.0 Appendices

AGN-242428 and AGN-231868 2012-201-005 – Statistical Analysis Plan (Stage 2) Version 1.0 – 07 December 2021

#### **Appendix A.** Protocol Deviations

According to ICH E3 2012 guideline, only important protocol deviations will be reported in CSR. The number and percentage of randomized participants with important protocol deviations will be summarized overall and by study intervention group for participants reported by protocol deviation categories:

- Participants who entered the study even though they did not satisfy the entry criteria
- Participants with inclusion criteria not met, overall and by inclusion criteria
- Participants with exclusion criteria met, overall and by exclusion criteria
- Participants developed withdrawal criteria during the study but were not withdrawn
- Participants received wrong treatment or incorrect dose of study treatment
- Participants took prohibited concomitant medication

#### **Appendix B.** Definition of Adverse Events of Special Interest

The following adverse events of special interest (AESI) (serious or nonserious) are defined in the protocol and will be summarized by PT terms listed in Table 5:

- AST and/or ALT increased to  $\geq$  5 ULN
- AST and/or ALT increased to ≥ 3 × ULN AND total bilirubin increased to ≥ 2 × ULN. Typically, all analytes will be obtained from the same sample, but they may come from multiple samples taken within a 24-hour period.
- AST and/or ALT increased to ≥ 3 × ULN with symptoms believed to be related to liver injury (e.g., fatigue, nausea, vomiting, right upper quadrant pain or tenderness or jaundice) or hypersensitivity (such as fever, rash, or eosinophilia > 5%)
- Potential Hy's Law cases:
  - o ALT and/or AST  $\geq$  3 × ULN AND
  - $\circ$  TBL  $\geq 2 \times$  ULN AND
  - $\circ$  Alkaline phosphatase  $< 2 \times ULN$

Table 5. List of Preferred Terms for Adverse Events of Special Interest

| Preferred Term (PT) | PT Code |
|--------------------------------------|----------|
| Aspartate aminotransferase increased | 10003481 |
| Alanine aminotransferase increased | 10001551 |
| Blood bilirubin increased | 10005364 |
| Blood alkaline phosphatase increased | 10059570 |

## Appendix C. Potentially Clinically Significant Criteria for Safety Endpoints

The potentially clinically significant criteria for clinical laboratory parameters, vital signs and ECG parameters are provided in the following sections.

Table 6. Potentially Clinically Significant Criteria for Clinical Laboratory Parameters

| Laboratory<br>Group | Parameter | SI Unit | PCS Low<br>Limit | PCS High<br>Limit |
|---|---|---|---|---|
| Hematology | Eosinophils absolute cell count | 10 <sup>9</sup> /L | _ | > 1.5 × ULN |
| | Hematocrit | % | < 0.8 × LLN | $\geq 1.2 \times ULN$ |
| | Hemoglobin | g/L | < 0.8 × LLN | $\geq 1.2 \times ULN$ |
| | Lymphocytes absolute cell count | 10 <sup>9</sup> /L | < 0.8 × LLN | > 1.2 × ULN |
| | Neutrophils absolute cell count | 10 <sup>9</sup> /L | < 0.6 × LLN | > 1.6 × ULN |
| | Platelet count (thrombocytes) | 10 <sup>9</sup> /L | < 0.5 × LLN | > 1.5 × ULN |
| | Red blood cell count | $10^{12}/L$ | < 0.8 × LLN | > 1.2 × ULN |
| | White blood cell count | 10 <sup>9</sup> /L | < 0.7 × LLN | > 1.8 × ULN |
| Chemistry | Alanine aminotransferase | U/L | | > 3 × ULN |
| | Albumin | g/L | < 0.9 × LLN | > 1.1 × ULN |
| | Alkaline phosphatase | U/L | | > 3 × ULN |
| | Aspartate aminotransferase | U/L | | > 3 × ULN |
| | Bilirubin, total | μmol/L | _ | > 1.5 × ULN |
| | Blood urea nitrogen | mmol/L | _ | > 1.3 × ULN |
| | Calcium | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| | Cholesterol, total | mmol/L | _ | > 1.2 × ULN |
| | Creatinine | μmol/L | _ | > 1.8 × ULN |
| | Glucose, fasting | mmol/L | < 0.8 × LLN | > 1.2 × ULN |
| | Glucose, nonfasting | mmol/L | < 0.8 × LLN | > 1.4 × ULN |
| | Phosphorus | mmol/L | < 0.8 × LLN | > 1.2 × ULN |
| | Potassium | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| | Protein, total | g/L | < 0.9 × LLN | > 1.1 × ULN |
| | Sodium | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| | Uric acid (urate) | μmol/L | | > 1.2 × ULN |

| Laboratory<br>Group | Parameter | SI Unit | PCS Low<br>Limit | PCS High<br>Limit |
|---|---|---|---|---|
| Urinalysis | Glucose | μmol/L | | ≥ 0.015 |
| | Glucose (alternate units) | _ | | ≥ 2+ |
| | рН | _ | < 0.9 × LLN | > 1.1 × ULN |
| | Protein | g/L | | ≥ 1.0 |
| | Protein (alternate units) | _ | | ≥ 2+ |
| | Specific gravity | _ | _ | > 1.1 × ULN |

LLN = lower limit of normal (value provided by the laboratory); PCS = potentially clinically significant; SI = *Le Système International d'Unités* (International System of Units); ULN = upper limit of normal (value provided by the laboratory)

Table 7. Potentially Clinically Significant Criteria for Vital Signs Parameters

| | | | PCS Criteria | |
|---|---|---|---|---|
| Parameter | Unit | PCS Category | Actual Value | Change from Baseline |
| Sitting Systolic BP | mmII.a | High | ≥ 180 | Increase of ≥ 20 |
| | mmHg | Low | ≤ 90 | Decrease of ≥ 20 |
| Sitting Diastolic BP | mmII.a | High | ≥ 105 | Increase of $\geq 15$ |
| | mmHg | Low | ≤ 50 | Decrease of ≥ 15 |
| Sitting Pulse rate | hom | High | ≥ 120 | Increase of $\geq 15$ |
| | bpm | Low | ≤ 50 | Decrease of ≥ 15 |
| Waight | kg | High | <del></del> | Increase of $\geq 7\%$ |
| Weight | | Low | <del></del> | Decrease of ≥ 7% |
| Dagninatam, Data | hom | High | ≥ 28 | _ |
| Respiratory Rate | bpm | Low | ≤ 8 | _ |
| Tommoroture | °C | High | > 38 | _ |
| Temperature | | Low | < 35 | _ |

BP = blood pressure; bpm = beats/breaths per minute

ECG values meeting *either* the actual value or change from baseline PCS high criteria will be categorized as PCS.



## Table 8. Potentially Clinically Significant Criteria for ECG Parameters

| Parameter | | PCS High Criteria | |
|--------------|------|-------------------|----------------------|
| | Unit | Actual Value | Change from Baseline |
| QRS interval | msec | ≥ 150 | _ |
| PR interval | msec | ≥ 250 | _ |
| QTcF | msec | > 500 | Increase > 60 |

QTcF = QTc Fridericia



## Appendix D. List of Abbreviations

| Abbreviation | Definition |
|--------------|----------------------------------------------|
| AE | adverse event |
| AESI | adverse event of special interest |
| AGN | Allergan |
| ATC | Anatomical therapeutic chemical |
| BCVA | best corrected visual acuity |
| CAE | controlled adverse environment |
| DED | dry eye disease |
| DMC | data monitoring committee |
| DMC | data monitoring committee |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| ETDRS | Early Treatment Diabetic Retinopathy Study |
| IOP | intraocular pressure |
| ITT | Intent-to-Treat |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NEI | National Eye Institute |
| ODS | Ocular Discomfort Scale |
| PCS | potentially clinically significant |
| PK | pharmacokinetic |
| PT | preferred term |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SOC | system organ class |
| TEAE | treatment-emergent adverse event |
| TESAE | treatment-emergent serious adverse event |
| WHO | World Health Organization |



### **Appendix E.** Changes to Protocol-planned Analyses

No statistical comparisons/tests among the study intervention groups will be performed for the safety data.

Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

## **Title Page**

#### **Protocol Title:**

A Multicenter, Vehicle-controlled, Double-Masked, Randomized Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Exploratory Efficacy of AGN-242428 and AGN-231868 in Participants with Dry Eye Disease

**Protocol Number:** 2012-201-005 [Stage 1]

Compound Number: AGN-242428 and AGN-231868

**Short Title:** 

Safety, Tolerability, Pharmacokinetics, and Efficacy of AGN-242428 and AGN-231868 in

Participants with Dry Eye Disease

Sponsor Name: Allergan Sales LLC

Legal Registered Address: 2525 Dupont Drive, Irvine, CA 92612, USA

**Regulatory Agency Identifier Number(s)** 

**Registry** ID

IND 139391, 139392



## **Table of Contents**

| Title Pag | Je | |
|------------|---------------------------------------|----|
| Table of | Contents | 2 |
| List of T | ables | 3 |
| SAP Vei | rsion History | 5 |
| 1. | Introduction | |
| 1.<br>1.1. | Objectives and Endpoints | |
| 1.2. | Study Design | |
| 2. | Statistical Hypotheses | 8 |
| 3. | Sample Size Determination | 9 |
| 4. | Analysis Sets | 10 |
| 5. | Statistical Analyses | 11 |
| 5.1. | General Considerations | |
| 5.2. | Participant Disposition. | 12 |
| 5.3. | Primary Endpoint(s) Analysis | |
| 5.4. | Secondary Endpoint(s) Analysis | 13 |
| 5.5. | | 13 |
| 5.6. | Safety Analyses | 13 |
| 5.6.1. | Extent of Exposure | 13 |
| 5.6.2. | Adverse Events | 14 |
| 5.6.2.1. | Adverse Events of Special Interest | 15 |
| 5.6.3. | Additional Safety Assessments | 16 |
| 5.6.3.1. | Clinical Laboratory Parameters | 16 |
| 5.6.3.2. | Potential Hy's Law | 17 |
| 5.6.3.3. | Vital Signs | 17 |
| 5.6.3.4. | Electrocardiogram | 18 |
| 5.6.3.5. | Physical Exam. | 19 |
| 5.6.3.6. | Best-corrected Visual Acuity | 19 |
| 5.6.3.7. | Intraocular Pressure | 20 |
| 5.6.3.8. | Biomicroscopy | 20 |
| 5.6.3.9. | Dilated Fundus Examination. | 21 |
| | Drop Tolerability Questionnaire Score | |
| 5.7. | Other Analyses | |
| 5.7.1. | Other Variables and/or Parameters | 22 |
| 5.7.1.1. | Pharmacokinetic Analyses | 22 |
| 5.7.2. | Subgroup Analyses | |
| 5.8. | Interim Analyses | 22 |
| 5.8.1. | Data Monitoring Committee | 22 |

## Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

| 6. | Supporting Documentation | 23 |
|---|---|---|
| 6.1. | Appendix 1: List of Abbreviations | |
| 6.2. | Appendix 2: Changes to Protocol-planned Analyses | |
| 6.3. | Appendix 3: Supporting Study Information | |
| 6.3.1. | 1. Demographics | |
| 6.3.2. | Baseline and Disease Characteristics | 27 |
| 6.3.3. | Protocol Deviations. | 27 |
| 6.3.4. | Medical and Ophthalmic History | |
| 6.3.5. | Prior/Concomitant Medications (Including Dictionary) | |
| 6.3.6. | Potentially Clinically Significant Criteria for Safety Endpoints | 28 |
| 6.3.6.1. | Potentially Clinically Significant Criteria for Clinical Laboratory | |
| (2.60 | Parameters | |
| 6.3.6.2. | Potentially Clinically Significant Criteria for Vital Signs | |
| 6.3.6.3.<br>6.4. | Potentially Clinically Significant Criteria for ECG Parameters | |
| 6.4.1. | Data Handling Conventions Study Intervention Conventions | |
| 6.4.1.1. | Analysis Days | |
| 6.4.1.2. | | |
| 6.4.1.3. | $\mathcal{I}$ | |
| 6.4.2. Repeated or Unscheduled Assessments | | |
| 6.4.3. | 1 | |
| 6.4.3.1. | Missing/Incomplete AE Start Date | 32 |
| 6.4.3.2. | Missing/Incomplete Medication Start Date | |
| 6.4.3.3. | Missing/Incomplete AE/Medication End Date | |
| 6.4.4. | Safety Endpoint Conventions | |
| 6.4.4.1. | Adverse Events | 33 |
| 7. | References | 32 |
| | List of Tables | |
| Table 1- | -1 Stage 1 Objectives | 6 |
| Table 4- | -1 Analysis Sets | 10 |
| Table 5- | -1 Statistical Methodology | 11 |
| Table 5- | -2 Participant Disposition Summaries | 13 |
| Table 5- | -3 Baseline Definitions | 13 |
| Table 5- | TEAE Summaries | 15 |
| Table 5- | Adverse Events of Special Interest | 16 |
| Table 5- | -6 Safety Laboratory Assessments | 16 |



## Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

| Table 5-7 | Clinical Laboratory Summaries | 17 |
|------------|------------------------------------------------------------|----|
| Table 5-8 | Potential Hy's Law Summaries | 17 |
| Table 5-9 | Vital Signs Summaries | 18 |
| Table 5-10 | Derivations of QTcF | 19 |
| Table 5-11 | ECG Summaries. | 19 |
| Table 5-12 | BCVA Summaries | 20 |
| Table 5-13 | IOP Summaries | 20 |
| Table 5-14 | Biomicroscopy | 21 |
| Table 5-15 | Dilated Fundus Examination. | 21 |
| Table 5-16 | Drop Tolerability Questionnaire Score | 21 |
| Table 6-1 | Abbreviations and Definitions of Terms. | 24 |
| Table 6-2 | Demographic Summaries | 27 |
| Table 6-3 | Baseline and Disease Characteristics Summaries | 27 |
| Table 6-4 | Medical History Summary | 28 |
| Table 6-5 | Clinical Laboratory PCS Criteria | 29 |
| Table 6-6 | Vital Sign PCS Criteria | 30 |
| Table 6-7 | ECG PCS Criteria | 30 |
| Table 6-8 | Analysis Day Definitions | 31 |
| Table 6-9 | Analysis Visit Definitions for Stage 1 | 31 |
| Table 6-10 | Imputation Scenarios | 32 |
| Table 6-11 | Initial Imputed Date Algorithm | 32 |
| Table 6-12 | Missing AE Severity and Relationship Imputation Algorithms | 33 |

Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

## **SAP Version History**

This Safety Statistical Analysis Plan (SAP) for Stage 1 of study 2012-201-005 is based on the protocol amendment 2, dated 27 April 2020.

| SAP Version History Summary | | | |
|---|---|---|---|
| SAP<br>Version | Approval<br>Date | Change | Rationale |
| 1 | | Not Applicable | Original version |
Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

### 1. Introduction

This SAP provides a technical and detailed elaboration of the statistical analyses of the Stage 1 safety data as outlined and specified in the final protocol of 2012-201-005 (Amendment 2, 27 April 2020). Specifications of tables and data listings are contained in a separate document. A separate SAP will be developed for Stage 2 data.

# 1.1. Objectives and Endpoints

#### Table 1-1 Stage 1 Objectives

| Stage 1 |
|---------------------|
| Primary Objectives: |

- To evaluate the safety and tolerability of up to three dose strengths of AGN-242428 and AGN-231868 and their respective vehicles in participants with dry eye disease (DED)
- To characterize the plasma and tear pharmacokinetics of AGN-242428 and AGN-231868 in participants with DED following a single bilateral administration; and 13 days of twice daily administration followed by a single administration to both eyes on the final day of administration

| Objective<br>Clinical<br>Category | Statistical<br>Category | Estimand/Variable |
|---|---|---|
| Safety | Primary | <ul> <li>Variables: Adverse events (AEs), clinical laboratory values, vital signs, electrocardiogram (ECG) findings, intraocular pressure (IOP), best-corrected visual acuity (BCVA), slit-lamp biomicroscopy, dilated fundus examination, Drop Tolerability Questionnaire score</li> <li>Population: Safety Population</li> <li>Analyses: Descriptive summary</li> </ul> |
| Pharmacokinetics <sup>a</sup> | Primary | <ul> <li>Variables: Systemic and tear pharmacokinetic parameters</li> <li>Following a single dose administration: area under the plasma or tear concentration versus time curve from time 0 to time of the last measurable concentration (AUC<sub>0-tlast</sub>) maximum plasma or tear drug concentration (C<sub>max</sub>), time of maximum plasma or tear drug concentration (T<sub>max</sub>), and terminal elimination half-life (t<sub>1/2</sub>)</li> <li>Following repeat dose administration: area under the plasma or tear concentration versus time curve from time 0 to the end of the dosing interval (AUC<sub>0-τ</sub>), C<sub>max</sub>, T<sub>max</sub>, minimum plasma or tear drug concentration at steady state (C<sub>min,ss</sub>), accumulation index (AI), and t<sub>1/2</sub></li> <li>Population: Pharmacokinetics population</li> <li>Analyses: Descriptive summary</li> </ul> |

Note: All estimand attributes explicitly identified for primary estimands only.

<sup>&</sup>lt;sup>a</sup> Analyses of Pharmacokinetics data will be described in a separate Pharmacokinetic Data Analysis Plan.

### Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

# 1.2. Study Design

Study 2012-201-005 is a Phase 1/2a, multicenter, vehicle-controlled, double-masked, randomized study conducted in 2 consecutive stages in participants with DED. Stage 1 will be conducted at 1 to 2 sites in the United States.

#### Stage 1

Stage 1 will evaluate the safety, tolerability, and pharmacokinetics (plasma and tear), of a maximum of 3 dose strengths of AGN-242428 ( ) and AGN-231868 ( ) in up to 3 consecutive cohorts (1A, 1B [high dose], and 1C [mid dose]) of participants with DED. There will be 24 participants in each cohort, with participants in each cohort randomized into 1 of 4 intervention arms:

- AGN-242428 (N = 9)
- AGN-231868 (N = 9)
- AGN-242428 vehicle (N = 3)
- AGN-231868 vehicle (N = 3)

All participants will receive 1 drop of the assigned intervention administered by the site staff to the left eye on Day 1 (Visit 2). In the absence of significant study intervention-related safety findings from this administration at the site, on Days 2 to 14, the participants will self-administer a single drop to both eyes, twice daily. On Day 15 (Visit 5), the participants will be administered a single drop to both eyes by the site staff.

The sponsor will decide whether to proceed to the next cohort after DMC review of safety data. If no significant safety or tolerability findings are identified in Cohort 1B, Cohort 1C will not be initiated.

#### Stage 2

Analysis of Stage 2 data will be discussed in a separate SAP.

No participant can be enrolled in more than 1 cohort and/or stage of the study.

If all doses are well tolerated, the duration of participation for each participant in the study will be as follows:

• For participants in Stage 1: approximately 1 month (Day -14 through collection of the last PK sample on Day 15)

# Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

# 2. Statistical Hypotheses

No hypothesis testing will be performed for Stage 1 safety data.

Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

# 3. Sample Size Determination

For Stage 1, the sample size is not based on statistical considerations and is determined empirically.

# Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

# 4. Analysis Sets

The analysis set for safety will consist of the population as defined below:

Table 4–1 Analysis Sets

| Population | Definition | Study Intervention |
|---|---|---|
| Safety | All participants who received at least one administration of | Actual received |
| | study intervention for stage 1 | |

Safety Statistical Analysis Plan

CONFIDENTIAL AGN-242428 AGN-231868 2012-201-005 [Stage 1]

# 5. Statistical Analyses

### **5.1.** General Considerations

The methodologies specified to individual variables are defined as follows:

Table 5-1 Statistical Methodology

| Methodology | Description |
|---|---|
| Categorical descriptives | <ul> <li>Number and percentage of participants in individual categories</li> <li>○ Participants with ≥ 1 qualifying event counted once per individual category</li> </ul> |
| PCS descriptives | <ul> <li>Number and percentage of participants meeting potentially clinically significant (PCS) criteria <ul> <li>○ Participants with ≥ 1 qualifying event counted once per PCS category</li> </ul> </li> <li>Percentage denominator = number of participants with available (non-missing) non-PCS baseline value(s) or available (non-missing) baseline and ≥1 non-missing postbaseline assessment</li> <li>○ Unevaluable assessments considered missing</li> </ul> |
| Continuous descriptives | <ul> <li>N1, mean, standard deviation (SD), Q1, Q3, median, minimum, maximum</li> <li>N1 = participants with non-missing value</li> </ul> |
| CFB descriptives | <ul> <li>Continuous descriptives for baseline, postbaseline, and change from baseline (CFB) values</li> <li>N1 = participants with non-missing values at both baseline and the specified postbaseline analysis by visit/timepoint</li> </ul> |
| Supportive data listing | <ul> <li>After table listings, i.e. the listing supports the findings from a table.</li> <li>Fully defined in the tables, figure, and listing specification document</li> </ul> |

CFB = change from baseline; PCS = potentially clinically significant; SD = standard deviation.

- An interim database lock will occur after completion of Stage 1. At the end of the study (completion of Stage 2), the final database lock will occur.
- All data will be provided in data listings which will be fully defined in the table, figure, and listing specification document. For these data listings, missing or incomplete dates or missing AE severity or relationship will be listed as is.
- The change from baseline values will be computed as the value for the post baseline visit minus the baseline value, unless otherwise indicated.
- Safety analyses will be based on the observed data. No imputation of missing values will be performed.

Safety Statistical Analysis Plan 2012-201-005 [Stage 1]

- Partial dates will be treated as missing in computations but will be listed in the data listings as they appear on the eCRFs unless otherwise specified. No imputation of missing values will be performed, unless otherwise specified.
- All statistical analysis will be performed using SAS version 9.4 or higher.
- MedDRA will be used to code adverse events and medical history.
- WHO Drug Dictionary will be used to code medications.
- Relative study day is defined as the number of days from the first dose date and will be presented in all data listings where a complete date is presented.
- The baseline for safety parameters will be the last assessment prior to the first administration of study intervention.
- Day 1 is the study day on which study intervention is first administered.
- The end of study for a participant is the last date that he/she participated in the study. The date will be captured on the end of intervention eCRF page.

# **5.2.** Participant Disposition

Number of participants screened for the study will be provided.

For each cohort, summary of study disposition will be provided by study intervention for the following:

- Number of participants randomized
- Number of participants treated
- Number of participants that completed the study
- Number of participants discontinued from the study
- eCRF-reported discontinuation reasons

In addition, a listing will be provided for participant disposition.

Safety Statistical Analysis Plan

CONFIDENTIAL AGN-242428 AGN-231868 2012-201-005 [Stage 1]

**Table 5-2** Participant Disposition Summaries

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Study disposition | Distribution in the Safety Population by study intervention for each cohort. | _ | Categorical<br>descriptives/<br>Supportive data<br>listing |

# 5.3. Primary Endpoint(s) Analysis

Not applicable.

# 5.4. Secondary Endpoint(s) Analysis

Not applicable.

# 5.5. Tertiary/Exploratory Endpoint(s) Analysis

Not applicable.

# **5.6.** Safety Analyses

Safety analyses will be based on the Safety Population.

Baseline assessments for applicable safety parameters are defined as follows:

**Table 5-3** Baseline Definitions

| Parameter | Baseline definition |
|---|---|
| <ul><li>Clinical laboratory evaluations</li><li>Vital signs</li><li>ECGs</li></ul> | Last non-missing assessment before the first dose for each participant in Stage 1 |
| • BCVA | |
| • IOP | |

# 5.6.1. Extent of Exposure

Exposure to the study treatment for the Safety Population will be summarized for treatment duration, calculated as last study intervention date - first study intervention date + 1. Descriptive statistics will be presented by cohort and study intervention group.

### Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

#### **5.6.2.** Adverse Events

An AE will be considered a TEAE if:

- The AE began on or after the first administration of study intervention, or
- The AE was present before the first administration of study intervention, but worsened (increased in severity or became serious) on or after the first dose of study intervention

An AE that occurs after the Exit or Early Termination visits will not be counted as a TEAE.

An AE will be considered a TESAE if it is a TEAE that additionally meets any SAE criterion.

TEAEs will be summarized by cohort and study intervention group using the Safety population.

If more than 1 AE is coded to the same preferred term for the same participant, the participant will be counted only once for that preferred term using the most severe and most related occurrence for the summarizations by severity and by relationship to study intervention.

Listings of all TEAEs, TESAEs, TEAEs leading to discontinuation by participant, and deaths will be presented.

AEs will be coded using MedDRA version 23.0 or newer. Unique participants reporting AEs in the following AE categories will be summarized by cohort and study intervention group for the Safety Population as follows:

Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

**Table 5-4 TEAE Summaries** 

| Parameters | Description | Methodology |
|---|---|---|
| AE | Overall summary by cohort and study intervention group only for the following categories: TEAEs Treatment-related TEAEs TESAEs Treatment-related TESAEs TEAEs leading to study discontinuation Deaths | Categorical descriptives |
| TEAEs | Overall summary by cohort and study intervention group and by SOC and PT Participants categorized overall and within each SOC and PT in decreasing frequency | Categorical descriptives |
| TEAEs by severity | Overall summary by cohort and study intervention group and by SOC, PT, and severity • Participants categorized overall and within each SOC and PT in decreasing frequency for the most severe occurrence | Categorical<br>descriptives |
| Treatment-related TEAEs | Overall summary by cohort and study intervention group and by SOC and PT Participants categorized overall and within each SOC and PT in decreasing frequency | Categorical descriptives |
| TESAEs | Overall summary by cohort and study intervention group and by SOC and PT <sup>a</sup> | Categorical<br>descriptives <sup>1</sup><br>Supportive data<br>listing |
| TEAEs leading to discontinuation | Overall summary by cohort and study intervention group and by SOC and PT <sup>a</sup> | Categorical<br>descriptives <sup>1</sup><br>Supportive data<br>listing |
| AESI | Overall summary by cohort and study intervention group and by SOC and PT <sup>a</sup> | Categorical<br>descriptives <sup>1</sup><br>Supportive data<br>listing |

<sup>&</sup>lt;sup>a</sup> Create summary tables only if at least 5 participants reported SAE, AEs leading to study discontinuation or AESI.

### **5.6.2.1.** Adverse Events of Special Interest

Any report of the following AESIs will be provided in a listing. A summary table will be created only if there are reports by at least 5 participants.

Safety Statistical Analysis Plan 2012-201-005 [Stage 1]

Table 5-5 Adverse Events of Special Interest

| Preferred Term (PT) | PT Code |
|--------------------------------------|----------|
| Aspartate aminotransferase increased | 10003481 |
| Alanine aminotransferase increased | 10001551 |
| Blood bilirubin increased | 10005364 |
| Blood alkaline phosphatase increased | 10059570 |

#### **5.6.3.** Additional Safety Assessments

#### **5.6.3.1.** Clinical Laboratory Parameters

**Table 5-6** Safety Laboratory Assessments

| Laboratory | | | |
|---|---|---|---|
| Assessments | · | | |
| Hematology | Platelet count | RBC indices: | WBC count with differential (absolute): |
| | RBC count | MCV | Neutrophils |
| | Hemoglobin | MCH | Lymphocytes |
| | Hematocrit | MCHC | Monocytes |
| | | | Eosinophils |
| | | | Basophils |
| Clinical Chemistry <sup>a</sup> | BUN | Potassium | Aspartate aminotransferase (AST) |
| | Creatinine | Sodium | Alanine aminotransferase (ALT) |
| | Glucose (fasting <sup>b</sup> ) | Calcium | Alkaline phosphatase |
| | Total protein | Cholesterol | Total, direct and indirect bilirubin |
| | Albumin | Chloride | |
| Routine Urinalysis | Specific gravity, pH, glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, | | |
| , | leukocyte esterase by dipstick | | |
| | Microscopic examination (if blood or protein is abnormal) | | |

<sup>&</sup>lt;sup>a</sup> In Stage 1, blood samples will be collected following 10-hour fasting period.

Descriptive statistics for quantitative clinical laboratory values (in SI units) at Screening, Exit visit, and changes from baseline at Exit/Early Termination visit will be presented by cohort and study intervention group for each clinical laboratory assessment.

Clinical laboratory test values will be considered PCS if they meet either the lower-limit or higher-limit PCS criteria listed in Table 6-5. The number and percentage of participants who have at least one PCS post-baseline clinical laboratory values will be tabulated by cohort and study intervention group at Exit visit. The percentages will be calculated based on the denominator of the number of participants with available non-PCS baseline values and at least one post-baseline value and the numerator of the number of participants with non-PCS baseline value and at least one PCS post-baseline-value.

<sup>&</sup>lt;sup>b</sup> Fasting requirement is for Stage 1 only

Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

A supportive listing of participants with postbaseline PCS values will be provided, including the participant number and baseline and postbaseline values, for the safety population. A listing of conversion factors to convert SI units to conventional units will be provided.

**Table 5-7** Clinical Laboratory Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| PCS values <sup>a</sup> | <ul> <li>Summary by laboratory category, laboratory test, and PCS criteria</li> <li>Participants with baseline PCS values excluded from analysis</li> <li>Parameters and PCS criteria specified in Sections 6.5.2.2 and 6.5.2.1, respectively</li> </ul> | Screening <sup>b</sup> , Exit <sup>c</sup> | PCS descriptives/<br>Supportive data<br>listing |
| Descriptives | Summary by laboratory category and laboratory test in SI and /or CV units and analysis visit Parameters specified in Section 6.5.2.2 | Screening <sup>b</sup> , Exit <sup>c</sup> | CFB descriptives |

<sup>&</sup>lt;sup>a</sup> Participants who report ≥ 1 postbaseline PCS value and all clinical laboratory for those participants will be listed.

#### 5.6.3.2. Potential Hy's Law

Potential Hy's Law criteria will be listed for the Safety Population as follows:

Table 5-8 Potential Hy's Law Summaries

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Potential Hy's Law<br>within 24-hour<br>window | Postbaseline assessment of the following laboratory parameters based on blood draws collected within a 24-hour period: • ALT or AST ≥ 3 × ULN • TBL ≥ 2 × ULN • ALP < 2 × ULN | Study Intervention<br>Period | Supportive data listing |

#### **5.6.3.3. Vital Signs**

Descriptive statistics for vital signs (systolic and diastolic blood pressures, pulse rate, weight, respiration rate, and temperature) at Screening, Baseline (Day 1) and changes from baseline values at each visit and at the Exit/Early Termination visit will be presented by cohort and study intervention group.

<sup>&</sup>lt;sup>b</sup> Visit will be used as baseline for change from baseline summaries.

<sup>&</sup>lt;sup>c</sup> Exit: Final or early termination visit.



Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

Vital sign values will be considered PCS if they meet either the lower-limit or higher-limit PCS criteria listed in Table 6-6. The number and percentage of participants who have at least one PCS post-baseline vital sign value will be tabulated by cohort and study intervention group. The percentages will be calculated based on the denominator of the number of participants with available baseline values or non-PCS baseline values (respiratory rate and temperature) and at least one post-baseline value and the numerator of the number of participants with non-PCS baseline value and at least one PCS post-baseline value.

A supportive listing of participants with postbaseline PCS values will be provided, including the participant number and baseline and postbaseline values, for the safety population.

**Table 5-9** Vital Signs Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| PCS values <sup>a</sup> | Summary by parameter and PCS criteria Denominator: available baseline or non-PCS baseline (respiratory rate or temperature) and at least one end-of-study or postbaseline values Parameters and PCS criteria specified in Sections 6.5.3.2 | Blood pressure, pulse rate, temperature: Day 1 <sup>b</sup> , Day 2, Day 8, Exit <sup>c</sup> Respiration rate, weight: Screening <sup>b</sup> , Exit <sup>c</sup> | PCS descriptives/ Supportive data listing <sup>a</sup> |
| Descriptives | and 6.5.3.1 respectively Summary by parameter and analysis visit Parameters specified in Section 6.5.3.2 | Blood pressure, pulse rate, temperature: Screening, Day 1 <sup>b</sup> , Day 2, Day 8, Exit <sup>c</sup> Respiration rate, weight: Screening <sup>b</sup> , Exit <sup>c</sup> | CFB descriptives |

<sup>&</sup>lt;sup>a</sup> Participants who report ≥ 1 postbaseline PCS value and all vital signs will be listed.

#### 5.6.3.4. Electrocardiogram

Descriptive statistics for ECG parameters (heart rate, RR interval, PR interval, QRS interval, QT interval, and QTc) at Baseline and Exit/Early Termination visits, and changes from baseline values at Exit/Early Termination visit will be presented by cohort and study intervention group.

The QTc will be calculated using the Fridericia correction (if the vendor does not provide). QTcF are derived as follows:

<sup>&</sup>lt;sup>b</sup> Visit will be used as baseline for change from baseline summaries.

<sup>&</sup>lt;sup>c</sup> Exit: Final or early termination visit.

Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

Table 5-10 Derivations of OTcF

| Parameter | Derivation if RR available | Derivation if RR unavailable |
|------------------|----------------------------|------------------------------|
| QTcF | QT | QT |
| (QTc Fridericia) | cubic root of RR | cubic root of 60/HR |

ECG parameter values will be considered PCS if they meet either the lower-limit or higher-limit PCS criteria listed in Table 6-7. The number and percentage of participants who have at least one PCS post-baseline ECG values will be tabulated for all participants by cohort and study intervention group. The percentages will be calculated based on the denominator of the number of participants with available non-PCS baseline values and at least one post-baseline value and the numerator of the number of participants with non-PCS baseline value and at least one PCS post-baseline value.

A supportive listing of participants with postbaseline PCS values will be provided, including the participant number and baseline and postbaseline values, for the safety population.

**Table 5-11 ECG Summaries** 

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| PCS values | Summary by parameter and PCS criteria Participants with baseline PCS values excluded from analysis Parameters and PCS criteria specified in Sections 6.5.4.2 and 6.5.4.3, respectively. | Screening <sup>b</sup> , Exit <sup>c</sup> | PCS<br>descriptives/<br>Supportive<br>data Listing <sup>a</sup> |
| Descriptives | Summary by parameter and analysis visit Parameters specified in Section 6.5.4.3 | Screening <sup>b</sup> , Exit <sup>c</sup> | CFB descriptives |

<sup>&</sup>lt;sup>a</sup> Participants who report ≥ 1 postbaseline PCS value and all ECG will be listed.

#### 5.6.3.5. Physical Exam

Abnormalities in PEs during Stage 1 of the study will be captured in medical history or AE data panels. Therefore, there will be no separate analyses for physical examination.

#### **5.6.3.6.** Best-corrected Visual Acuity

BCVA will be measured in each eye using the ETDRS chart. Descriptive statistics for BCVA at Screening, Baseline (Day 1), and changes from baseline at each postbaseline visit will be presented by cohort, and study intervention group for each eye. Vision loss will also be

<sup>&</sup>lt;sup>b</sup> Visit will be used as baseline for change from baseline summaries.

<sup>&</sup>lt;sup>c</sup> Exit: Final or early termination visit.

#### Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

summarized by study intervention group for each eye at each visit in a categorical tabulation as severe ( $\geq$  30 letters decrease from baseline), moderate ( $\geq$  15 and < 30 letters decrease from baseline) and no loss or mild (< 15 letters decrease from baseline).

Table 5-12 BCVA Summaries

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Vision loss | <ul> <li>Severe vision loss</li> <li>(&gt;= 30 letters decrease from baseline)</li> <li>Moderate vision loss</li> <li>(&gt;= 15 and &lt; 30 letters decrease from baseline)</li> <li>No loss or mild vision loss</li> <li>(&lt;15 letters decrease from baseline)</li> </ul> | Treatment Period | Categorical descriptives |
| BCVA | Raw values and change from baseline | Treatment Period | CFB descriptives |

#### 5.6.3.7. Intraocular Pressure

IOP will be measured in each eye using the Goldmann applanation tonometer. At least 2 measurements will be taken for each eye. If the 2 independent measurements differ by  $\leq$  2 mm Hg, a third measurement is not required, and the 2 measurements will be recorded. If the first 2 measurements differ by > 2 mm Hg, a third measurement must be made, and all 3 measurements will be recorded. The mean of the 2 (or 3) measures will be used as the IOP value. If, for any reason, only a single measurement is obtained, then this measurement will be used as the IOP value.

Descriptive statistics for IOP at Screening, Baseline (Day 1), and changes from baseline and number of participants reporting IOP > 21 mm Hg at each postbaseline visit will be presented by cohort and study intervention group for each eye.

**Table 5-13 IOP Summaries** 

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| IOP category | IOP > 21 mmHg (raw value) | Treatment period | Categorical descriptives |
| IOP | Raw values and change from baseline | Treatment period | CFB descriptives |

#### 5.6.3.8. Biomicroscopy

Slit-lamp biomicroscopy exam will be performed in each eye.

The number of participants with biomicroscopy findings of any severity increase from baseline at one or more visits will be generated for each MedDRA preferred terms by cohort and study

#### Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

intervention group for each eye. For findings under "other pathology" which are not associated with a severity grade, a status change from absent to present will be treated as an increase of severity in the analysis.

Table 5-14 Biomicroscopy

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Biomicroscopy | Any severity increase from baseline for each eye | Treatment period | Categorical descriptives |

#### **5.6.3.9.** Dilated Fundus Examination

Lens, vitreous, fundus, and optic nerve will be evaluated for pathology. If pathology is present, it will be recorded.

Cup/disc ratio will be reported using 0.0 to 1.0 scale according to an Armaly chart. Lens status will be assessed as phakic, pseudophakic, or aphakic. Cataract assessment for presence and severity of nuclear, cortical and posterior subcapsular cataract lens opacities will be evaluated. Each type of cataract severity and change from baseline will be evaluated. These data will be presented as listings only.

Table 5-15 Dilated Fundus Examination

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Dilated Fundus<br>Examination | Listing for the following data: Cup/disc ratio Lens status Cataract assessment | Treatment period | Listing |

### **5.6.3.10. Drop Tolerability Questionnaire Score**

Participants will be asked to rate the acute overall tolerability attributes of study interventions on an 8-question VAS Drop Tolerability Questionnaire. Descriptive statistics for each question at Baseline (Day 1), and changes from baseline at each postbaseline visit will be presented by cohort and study intervention group.

Table 5-16 Drop Tolerability Questionnaire Score

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Drop Tolerability Questionnaire VAS | Raw values and change from baseline | Treatment period | CFB descriptives |
| score | | | |

Safety Statistical Analysis Plan 2012-201-005 [Stage 1]

### 5.7. Other Analyses

#### 5.7.1. Other Variables and/or Parameters

#### **5.7.1.1.** Pharmacokinetic Analyses

Pharmacokinetic blood and tear (both eyes) sampling times and plasma and tear concentrations of AGN-242428 and AGN-231868 will be listed for the Safety Population. PK analyses will be described in the PK data analysis plan.

### 5.7.2. Subgroup Analyses

No subgroup analysis is planned for this study.

### 5.8. Interim Analyses

There is no interim analysis planned.

There are 2 database locks planned. The first database lock will take place after completion of Stage 1. At this time, the data for Stage 1 will be unmasked and topline data analyses will be performed. A topline report will be created in lieu of an interim CSR.

#### **5.8.1.** Data Monitoring Committee

The DMC will be composed of the sponsor's internal members who will be masked to the interventions. However, data can be unmasked at the DMC's discretion at any time.

In Stage 1, at the end of each cohort, the DMC will review the safety data and provide a recommendation on whether the study can proceed to the next cohort. In Stage 1, it is possible that only 1 of the interventions will proceed to the next cohort and/or to Stage 2.

All details of the committee membership, procedures for safety review, frequency of review, and communication between the safety review committee and other information will be detailed in the DMC charter

# Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

# **6.** Supporting Documentation

Additional study population, baseline characteristics, and pre-defined safety criteria can be found in Section 6.3.

Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

# **6.1.** Appendix 1: List of Abbreviations

### Table 6-1 Abbreviations and Definitions of Terms

| Abbreviation/Term | Definition |
|---|---|
| AE | adverse event |
| AESI | adverse event of special interest |
| AI | accumulation index |
| ALT | alanine aminotransferase |
| AST | aspartate aminotransferase |
| ALP | alkaline phosphatase |
| AUC | area under the curve |
| AUC0-tlast | area under the plasma or tear concentration versus time curve from time 0 to time of the last measurable concentration |
| ΑUC0-τ | area under the plasma or tear concentration versus time curve from time 0 to the end of the dosing interval |
| BCVA | best-corrected visual acuity |
| BID | twice daily |
| BP | Blood pressure |
| bpm | beats/breaths per minute |
| BUN | blood urea nitrogen |
| CAE | controlled adverse environment |
| CFB | change from baseline |
| Cmax | maximum plasma or tear drug concentration |
| Cmin,ss | minimum plasma or tear drug concentration at steady state |
| CRF | case report form |
| CSR | Clinical Study Report |
| DED | dry eye disease |
| DMC | data monitoring committee |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| ETDRS | Early Treatment Diabetic Retinopathy Study |
| FDA | Food and Drug Administration |
| hCG | human chorionic gonadotropin |
| ICH | International Council on Harmonization |
| IND | investigational new drug |
| IOP | intra-ocular pressure |
| LD | last day of the month |
| LLN | lower limit of normal |
| MedDRA | Medication Dictionary for Regulatory Activities |
| MCV | mean corpuscular volume |
| MCH | mean corpuscular hemoglobin |
| MCHC | mean corpuscular hemoglobin concentration |
| MM | available start date month |

# Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

| Abbreviation/Term | Definition |
|---|---|
| MSP | medical safety physician |
| NA | not applicable |
| OD | right eye |
| OS | left eye |
| OTC | over-the-counter |
| PE | physical examination |
| PCS | potentially clinically significant |
| PK | pharmacokinetic |
| PT | Preferred Term |
| QTc | QT Interval Corrected for Heart Rate |
| QTcF | QT Interval Corrected for Heart Rate Using the Fridericia Formula $(Qtcf = QT/(RR)^{1/3})$ |
| RBC | red blood cell |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SAS | Statistical Analysis System |
| SD | Standard deviation |
| SI | Le Système International d'Unités (International System of Units) |
| SOC | System Organ Class |
| SoA | schedule of activities |
| t <sub>1/2</sub> | terminal elimination half-life |
| TBL | total bilirubin |
| TEAE | treatment-emergent adverse event |
| TESAE | treatment-emergent serious adverse event |
| THC | tetrahydrocannabinol |
| ULN | upper limit of normal |
| WBC | white blood cell |
| WHO | World Health Organization |
| WOCBP | woman of childbearing potential |
| YYYY | available start date year |

Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

# 6.2. Appendix 2: Changes to Protocol-planned Analyses

There are no changes from the protocol-planned analyses.

# 6.3. Appendix 3: Supporting Study Information

### 6.3.1. Demographics

Demographics will be summarized descriptively by cohort and study intervention group for the Safety Population, as follows:

Table 6-2 Demographic Summaries

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Age | Age (years) | _ | Categorical descriptives |
| Sex, race, and ethnicity | eCRF categories | _ | Categorical descriptives |

Demographic and baseline characteristics will be provided in a listing.

#### 6.3.2. Baseline and Disease Characteristics

Baseline characteristics will be summarized descriptively by cohort and study intervention group for each eye for the Safety Population as follows:

Table 6-3 Baseline and Disease Characteristics Summaries

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Baseline characteristics | <ul> <li>Height (m)</li> <li>Weight (kg)</li> <li>Body mass index (BMI)</li> <li>Weight (kg) / height (m)<sup>2</sup></li> </ul> | Last assessment<br>before the first dose<br>date of the study<br>intervention | Continuous<br>descriptives |
| Disease characteristics | • BCVA | Last assessment<br>before the first dose<br>of the study<br>intervention<br>[Screening, Day 1] | Continuous<br>descriptives |

#### 6.3.3. Protocol Deviations

A data listing of any significant protocol deviations will be provided for the Safety Population.

#### 6.3.4. Medical and Ophthalmic History

Participants' medical and ophthalmic history, encompassing abnormalities and surgeries data, will be coded using the MedDRA, version 23.0 or higher. Reported medical events, ophthalmic

### Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

events and surgical history will be summarized using MedDRA SOC and PT by cohort and study intervention group for the Safety Population. Medical history includes prior medical history (prior to Day 1, first dose date) and still ongoing.

Table 6-4 Medical History Summary

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Medical history | Abnormalities and surgeries | _ | Categorical descriptives |
| Ophthalmic history | Abnormalities and surgeries | _ | Categorical descriptives |

SOCs will be sorted alphabetically; PTs will be sorted in descending frequency in the highest dose strength group.

### 6.3.5. Prior/Concomitant Medications (Including Dictionary)

The medication data will be coded using the WHO Drug Dictionary Enhanced, version MAR 2017 or newer. Prior medication is defined as any medication taken prior to the start of study intervention regardless of stop date of the medication. Concomitant medication is defined as any medication taken after the start of study intervention regardless of the start date of the medication.

Prior and concomitant medications will be coded using the Anatomical Therapeutic Chemical code (4th level, or most specific level available if 4th level is unavailable).

Medications data along with prior or concomitant medication flag will be listed for the Safety Population.

#### 6.3.6. Potentially Clinically Significant Criteria for Safety Endpoints

The potentially clinically significant criteria for clinical laboratory parameters, vital signs, and ECG parameters are provided in the following sections.



2012-201-005 [Stage 1]

# 6.3.6.1. Potentially Clinically Significant Criteria for Clinical Laboratory Parameters

Laboratory assessments values meeting any of the following PCS low or PCS high criteria will be categorized as PCS:

Table 6-5 Clinical Laboratory PCS Criteria

| Laboratory<br>Group | Parameter | SI Unit | PCS Low<br>Limit | PCS High<br>Limit |
|---|---|---|---|---|
| Hematology | Eosinophils absolute cell count | 10 <sup>9</sup> /L | _ | > 1.5 × ULN |
| | Hematocrit | % | < 0.8 × LLN | ≥ 1.2 × ULN |
| | Hemoglobin | g/L | < 0.8 × LLN | ≥ 1.2 × ULN |
| | Lymphocytes absolute cell count | 10 <sup>9</sup> /L | < 0.8 × LLN | > 1.2 × ULN |
| | Neutrophils absolute cell count | 10 <sup>9</sup> /L | < 0.6 × LLN | > 1.6 × ULN |
| | Platelet count (thrombocytes) | 10 <sup>9</sup> /L | < 0.5 × LLN | > 1.5 × ULN |
| | Red blood cell count | $10^{12}/L$ | < 0.8 × LLN | > 1.2 × ULN |
| | White blood cell count | 10 <sup>9</sup> /L | < 0.7 × LLN | > 1.8 × ULN |
| Chemistry | Alanine aminotransferase | U/L | _ | > 3 × ULN |
| | Albumin | g/L | < 0.9 × LLN | > 1.1 × ULN |
| | Alkaline phosphatase | U/L | _ | > 3 × ULN |
| | Aspartate aminotransferase | U/L | _ | > 3 × ULN |
| | Bilirubin, total | μmol/L | _ | > 1.5 × ULN |
| | Blood urea nitrogen | mmol/L | _ | > 1.3 × ULN |
| | Calcium | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| | Cholesterol, total | mmol/L | _ | > 1.2 × ULN |
| | Creatinine | μmol/L | _ | > 1.8 × ULN |
| | Glucose, fasting | mmol/L | < 0.8 × LLN | > 1.2 × ULN |
| | Glucose, nonfasting | mmol/L | < 0.8 × LLN | > 1.4 × ULN |
| | Phosphorus | mmol/L | < 0.8 × LLN | > 1.2 × ULN |
| | Potassium | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| | Protein, total | g/L | < 0.9 × LLN | > 1.1 × ULN |
| | Sodium | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| | Uric acid (urate) | μmol/L | _ | > 1.2 × ULN |
| Urinalysis | Glucose | μmol/L | _ | ≥ 0.015 |
| | Glucose (alternate units) | _ | _ | ≥ 2+ |
| | рН | _ | < 0.9 × LLN | > 1.1 × ULN |
| | Protein | g/L | | ≥ 1.0 |
| | Protein (alternate units) | _ | | ≥ 2+ |
| | Specific gravity | | | > 1.1 × ULN |

Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

### 6.3.6.2. Potentially Clinically Significant Criteria for Vital Signs

Vital sign values meeting *both* the actual value and change from baseline PCS criteria will be categorized as PCS:

Table 6-6 Vital Sign PCS Criteria

| | | | PCS Criteria | |
|---|---|---|---|---|
| Parameter | Unit | PCS Category | Actual Value | Change from Baseline |
| Sitting Systolic BP | mmHg | High | ≥ 180 | Increase of $\geq 20$ |
| | | Low | ≤ 90 | Decrease of $\geq 20$ |
| Sitting Diastolic BP | mmHg | High | ≥ 105 | Increase of $\geq 15$ |
| | | Low | ≤ 50 | Decrease of $\geq 15$ |
| Sitting Pulse rate | bpm | High | ≥ 120 | Increase of $\geq 15$ |
| | | Low | ≤ 50 | Decrease of $\geq 15$ |
| Weight | kg | High | <del></del> | Increase of $\geq 7\%$ |
| weight | | Low | <del></del> | Decrease of ≥ 7% |
| Dagnington: Data | bpm | High | ≥ 28 | _ |
| Respiratory Rate | | Low | ≤ 8 | |
| Tommoreture | °C | High | > 38 | _ |
| Temperature | | Low | < 35 | _ |

### 6.3.6.3. Potentially Clinically Significant Criteria for ECG Parameters

ECG values meeting *either* the actual value or change from baseline PCS high criteria will be categorized as PCS:

Table 6-7 ECG PCS Criteria

| | | PCS High Criteria | |
|--------------|------|-------------------|----------------------|
| Parameter | Unit | Actual Value | Change from Baseline |
| QRS interval | msec | ≥ 150 | _ |
| PR interval | msec | ≥ 250 | _ |
| QTcF | msec | > 500 | Increase > 60 |

Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

# **6.4.** Data Handling Conventions

### **6.4.1.** Study Intervention Conventions

### 6.4.1.1. Analysis Days

Study days are defined as follows:

Table 6-8 Analysis Day Definitions

| Term | Description |
|---|---|
| Study Day | Relative to study intervention start date If analysis date ≥ intervention start date: |
| | <ul> <li>Day = analysis date - study intervention start date + 1</li> <li>Day 1 = study intervention start date</li> </ul> |
| | If analysis date < intervention start date: • Day = analysis date - study intervention start date • Day -1 = day before study intervention start date |
| | o There is no Day 0 |

### 6.4.1.2. Analysis Window

Table 6-9 Analysis Visit Definitions for Stage 1

| Scheduled Visit | Target Day of the<br>Visit | Analysis Visit Window |
|------------------|----------------------------|--------------------------|
| Visit 2/Baseline | Day 1 | Day 1 |
| Visit 3 | Day 2 | Days [2, 5] |
| Visit 4 | Day 8 | Days [6, 11] |
| Visit 5 | Day 15 | Day 12 to study exit day |

### 6.4.1.3. Missing/Incomplete Intervention End Date

If the investigator is unable to provide the study intervention end date, study intervention end date will be imputed to the last available dosing record date.

#### **6.4.2.** Repeated or Unscheduled Assessments

If postbaseline assessments are repeated or if unscheduled assessments occur, the last postbaseline assessment will be used as the postbaseline assessment for generating summary statistics. However, all postbaseline assessments will be used for PCS value determinations, and all assessments will be presented in the supportive data listings.

Safety Statistical Analysis Plan 2012

2012-201-005 [Stage 1]

#### 6.4.3. Missing Date Imputation

Dates may be imputed with year, month, and day values under certain scenarios:

**Table 6-10** Imputation Scenarios

| | | Complete | | |
|----------|------|----------|-----|-----------|
| Scenario | Year | Month | Day | Imputable |
| 1 | Yes | Yes | Yes | Complete |
| 2 | Yes | Yes | _ | Yes |
| 3 | Yes | _ | Yes | Noa |
| 4 | Yes | _ | _ | Yes |
| 5 | _ | Yes | Yes | Noa |
| 6 | _ | Yes | _ | Noa |
| 7 | _ | _ | Yes | Noa |
| 8 | _ | _ | _ | Yes |

<sup>&</sup>lt;sup>a</sup> Not allowed per database design.

Dates will be imputed initially toward a specified target date for imputable scenarios 2, 4, and 8, and adjusted against the latest reasonable dates. The initial imputed date is determined by the following algorithm:

Table 6-11 Initial Imputed Date Algorithm

| Available Year | | Available Month (MM) | | |
|---|---|---|---|---|
| (YYYY) | Missing | < Target Month | = Target Month | > Target Month |
| Missing | Target Date | | _ | |
| < Target Year | YYYY-12-31 | | YYYY-MM-LD | |
| = Target Year | Target Date | YYYY-MM-LD | Target Date | YYYY-MM-01 |
| > Target Year | YYYY-01-01 | | YYYY-MM-01 | |

#### 6.4.3.1. Missing/Incomplete AE Start Date

Imputation of dates with missing day and/or month is only applied to TEAEs. If adequate information is available, no imputation is needed. TEAE start dates with missing day or month will be imputed as following:

- If day and month are missing but year is available, then the imputed day and month will be 01 Jan or the initial study intervention administration date if they have the same year, whichever is later (because TEAE onset is not expected prior to administration of study intervention)
- If day is missing but the month and year are available, then the imputed day will be the first day of the month or the initial injection date if they have the same month and year, whichever is later.

### Safety Statistical Analysis Plan

2012-201-005 [Stage 1]

### 6.4.3.2. Missing/Incomplete Medication Start Date

Medication start dates will be imputed as the minimum of the following:

- Initial imputed date, where target date = Treatment start date -1
- Complete end date

### 6.4.3.3. Missing/Incomplete AE/Medication End Date

Imputation of dates with missing day and/or month is only applied to TEAEs when AE duration is calculated. If adequate information is available, no imputation is needed. TEAE end dates with missing day or month will be imputed as following:

• If day and month are missing but year is available, then the imputed day and month will be 31 Dec or the study exit date if they have the same year, whichever is earlier

If day is missing but the month and year are available, then the imputed day will be the last day of the month or the study exit date if they have the same month and year, whichever is earlier.

### **6.4.4.** Safety Endpoint Conventions

#### 6.4.4.1. Adverse Events

#### **6.4.4.1.1.** Missing Intensity or Relationship

If the investigator is unable to provide the actual values, the following imputations will be applied:

Table 6-12 Missing AE Severity and Relationship Imputation Algorithms

| Missing Value | Imputation | Timing |
|---------------|------------|----------------------------------------|
| Severity | Mild | AEs before the first dose of the study |
| | | intervention in the study |
| | Severe | AEs on or after the first dose of the |
| | | study intervention in the study |
| Relationship | NA | AEs before the first dose of the study |
| | | intervention in the study |
| | Related | AEs on or after the first dose of the |
| | | study intervention in the study |

Safety Statistical Analysis Plan 2012

2012-201-005 [Stage 1]

# 7. References

Not applicable.